CLINICAL TRIAL: NCT03677063
Title: Usefulness of Sterile Adhesive Dressing at the Exit-site of Peritoneal Dialysis Catheter: a Pilot Study
Brief Title: Usefulness of Sterile Adhesive Dressing at the Exit-site of Peritoneal Dialysis Catheter
Acronym: PANCADIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A00379-46
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2022-02

CONDITIONS: Peritoneal Dialysis
Keywords: peritoneal dialysis; dressing; exit-site; catheter; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dressing (No Intervention): It is the historical cohort which is composed of patients over 18 years of age treated by peritoneal dialysis in the nephrology department of Universty Hospital of Caen Normandie. Patients with the same non-inclusion criteria as the experimental group will not be included. The data will be extracted from the Registry of Peritoneal Dialysis of French Language. The number of patients included from the register can not be fixed in advance; this number will correspond to the 4-year follow-up at the start date of the study to ensure at least two years of patient follow-up
  Usually care
  First dressing 5 or 10 days after the pose of the catheter :
  * Cleaning emergence with antiseptic soap
  * Rinsing with saline
  * Drying
  * Application of a hazelnut mupirocin on the exit-site
  * Application of an occlusive dressing on the exit-site Then, care is the same. Exit-site care is performed daily if the patient takes a shower or twice a week.
- No dressing (Experimental): No application of sterile dressing at the exit-site of periotoneal dialysis catheter for all patients (30 days after the placement of the peritoneal dialysis catheter)
  Interventions: Other: No dressing

INTERVENTIONS:
Other: No dressing — Then, care is the same and exit-site remains covered with an occlusive dressing to promote tunnel epithelialization and healing. The shower is forbidden during this period.
  Arms: No dressing

SUMMARY:
Infection of peritoneal dialysis fluid is a major complication in patients treated with peritoneal dialysis (PD). The aim of catheter emergence care is to reduce bacterial contamination of the peritoneum. The recommendations of the International Society of Peritoneal Dialysis do not provide information on the frequency of care delivery or the usefulness of a sterile adhesive dressing. Thus each treatment center applies a protocol of its own. Dressing is common practice although its safety and interest are not demonstrated.

The usefulness of dressing is still to be demonstrated. On the other hand, the efficacy of the application in prevention of a cream of mupirocin at emergence on the reduction of the risk of infection with staphylococcus aureus (SA), the most frequent germ found in peritonitis, has been demonstrated. A Spanish study showed that during a peritoneal infection at SA the site most frequently colonized by a similar strain of SA was the emergence of the catheter.

It can be considered that an infection of the dialysis liquid in PD is not only related to the quality of emergency care but also to manipulations during exchanges.

Given the number of patients involved in PD in France, it is difficult to obtain sufficient power to formally demonstrate the non-inferiority of the absence of dressing.

Therefore, the investigators propose a descriptive, exploratory study of events that may occur in PD when a dressing is not applied. This is a step prior to performing a multicenter randomized comparative study that will aim to show the non-inferiority of the absence of dressing compared to the application of a dressing on the incidence of fluid infection. peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* patient who has been informed and has given free and informed consent
* patient affiliated to a social security scheme

Exclusion Criteria:

* inclusion of the patient in another biomedical research protocol that influences the risk of infection
* burial of the catheter before the initiation of dialysis treatment second attempt at treatment with peritoneal dialysis following catheter removal and resection
* patient under curatorq
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Infectious event | 24 months
  Time until the occurrence of an infectious event:
  * Infection of Staphylococcus aureus peritoneal dialysis fluid (SA) within 24 months of follow-up
  * Infection of peritoneal dialysis fluid other than AS within 24 months of follow-up
  * Emergence infection during 24 months of follow-up
  * Peritonitis at SA and simultaneous presence of SA at emergence within 24 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: SONIA GUILLOUET, PhD's, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided